CLINICAL TRIAL: NCT05758259
Title: The Efficacy and Safety of Topical Vitamin D and Supplementation In Acne Vulgaris The Study of VDR, IL-1β, IL-6, IL-10 and IL-17 Expression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Nelly Herfina Dahlan Sp.KK, M.Kes, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KET-922/2022
Record Dates: First submitted 2023-01-08; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Acne Vulgaris; Vitamin D
MeSH Terms: conditions — Acne Vulgaris | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- combination vitamin D oral and topical cholecalciferol (Experimental): combination topical vitamin D and supplementation Daily supplementation (1x/day, in the morning) and topical application (2x/day, in the morning and in the afternoon, minimum duration 4 hours on the skin) for 56 days Daily supplementation (1x/day, in the morning) and topical application (2x/day, in the morning and in the afternoon, minimum duration 4 hours on the skin) for 56 days
  Interventions: Drug: combination oral and topical vitamin D
- oral placebo and topical vitamin D (Active Comparator): oral placebo and topical vitamin D Daily supplementation (1x/day, in the morning) and topical application (2x/day, in the morning and in the afternoon, minimum duration 4 hours on the skin) for 56 days
  Interventions: Drug: oral placebo and topical cholecalciferol
- oral placebo and basic ingredient placebo topical vitamin D (Placebo Comparator): Daily supplementation (1x/day, in the morning) and topical application (2x/day, in the morning and in the afternoon, minimum duration 4 hours on the skin) for 56 days
  Interventions: Drug: oral placebo and basic ingredient placebo topical vitamin D

INTERVENTIONS:
Drug: combination oral and topical vitamin D — combination vitamin D 2000 IU 1x1 and topical 7-Dehydrocholesterol 5000 mcg 2x1
  Arms: combination vitamin D oral and topical cholecalciferol
Drug: oral placebo and topical cholecalciferol — oral placebo and topical 7-Dehydrocholesterol 5000 mcg 2x1
  Arms: oral placebo and topical vitamin D
Drug: oral placebo and basic ingredient placebo topical vitamin D — oral placebo and basic ingredient placebo topical vitamin D similar to the ointment
  Arms: oral placebo and basic ingredient placebo topical vitamin D

SUMMARY:
Introduction This document is a clinical trial protocol. This research will be conducted based on the standards of the Good Clinical Trial Method and regulations from the relevant institutions and ethics committees.

Background Acne vulgaris (AV) is a chronic inflammatory disease with multifactorial causes in the skin's pilosebaceous follicular units, with clinical manifestations in the form of comedones, papules, pustules, nodes, and pseudocysts. The following factors are considered important for the etiology of AV: increased rate of sebum excretion, endocrinological factors such as androgens, abnormal keratinization of the follicular infundibulum, the proliferation of Cutibacterium acnes (C. acnes), and inflammation. Recent studies at the molecular and cellular levels have clarified how these factors interact and the role of the innate immune system. Inflammatory processes have been demonstrated in all types of lesions - preclinical microcomedones, comedones, inflammatory lesions, 'post inflammatory' erythema or hyperpigmentation, and scarring. Inflammation localized to the pilosebaceous can be considered a hallmark of acne and should be managed through several therapeutic routes. Clinicians tend to think that oral antibiotics should be used to treat inflammation in acne. However, this treatment are associated with resistance and low outcome due to its adverse events such as erythema, desquamation, and dry skin. There is evidence of the use and opportunity of vitamin D as a novelty treatment influencing the immune system. 25OHD and 1,25(OH)2D are both catabolized by CYP24A1. 1,25(OH)2D is a ligand for the vitamin D receptor (VDR), a transcription factor that binds to sites in DNA called vitamin D response elements (VDRE). Thousands of these binding sites regulate hundreds of genes through several signaling pathways in different cell types, including their regulation in immune cells by toll-like receptors (TLRs), the primary signaling nucleus of C. acnes that interacts with the innate immune system, causing acute and chronic inflammation.

Study Objectives Primary Objective The primary objective of this study is to evaluate the efficacy and safety of combination topical vitamin D and supplementation as adjuvant therapy in acne vulgaris compared to placebo and topical vitamin D monotherapy.

Secondary Objective(s) To assess Vitamin D Receptor (VDR) expression on acne lesion and blood sample To assess the effect of combination topical vitamin D and supplementation on IL-1β expression on acne lesion To assess the effect of combination topical vitamin D and supplementation on IL-6 expression on acne lesion To assess the effect of combination topical vitamin D and supplementation on IL-10 expression on acne lesion To assess the effect of combination topical vitamin D and supplementation on IL-17 expression on acne lesion

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with moderate or severe acne vulgaris
* Aged over 18-50 years.
* During the study, were willing not to use skin care products either in oral and/or topical form on the face, as well as other treatments outside of standard AV treatment.
* Willing to take part in the examination and treatment in accordance with the provisions of the study and follow the control time schedule in accordance with the predetermined research plan also willing to sign the informed consent form.

Exclusion Criteria:

* Women who are pregnant and breastfeeding.
* Have history using topical antibiotics in the past 2 weeks.
* Have history using topical corticosteroids in the past 2 weeks.
* Have history taking vitamin D supplements in the last 1 month.
* Have history taking oral antibiotics in the last 1 month.
* Have history using oral corticosteroid use in the last 1 month.
* Have history using oral and topical retinoid use in the last 3 months.
* Have history using topical BPO in the last 1 month.
* Using hormonal contraception for women.
* Have history of drug allergies or skin disorders due to side effects of first-line therapy drugs for moderate/severe acne vulgaris.
* Impaired liver and kidney function.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | baseline and week 8th
  Changes in counts of inflammation and non-inflammation lesions (assessed in week 8th)
Existence in VDR expression on acne lesion | baseline
  VDR count on CD 45 flowcytometry
Changes from baseline in IL-1β expression on acne lesion | baseline and week 8th
  IL-1β expression in pg/mL
Changes from baseline in IL-6 expression on acne lesion | baseline and week 8th
  IL-6 expression in pg/mL
Changes from baseline in IL-10 expression on acne lesion | baseline and week 8th
  IL-10 expression in pg/mL
Changes from baseline in IL-17 expression on acne lesion | baseline and week 8th
  IL-17 expression in pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Derived] Dahlan NH, Sitohang IBS, Indriatmi W, Wibowo H, Enggy LE. Correlation Between Reduced IL-1beta Levels in Acne Lesions and the Decrease in Acne Inflammatory Lesions Following Topical Vitamin D Administration: A Double-Blind Randomized Controlled Trial. Clin Cosmet Investig Dermatol. 2024 Oct 1;17:2183-2195. doi: 10.2147/CCID.S475068. eCollection 2024. PMID 39372262

DOCUMENTS (1):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT05758259/Prot_000.pdf